CLINICAL TRIAL: NCT02086461
Title: Pylorus Dysfunction After Esophagectomy. Effect of Pneumatic Dilatation.
Brief Title: Pylorus Dysfunction After Esophagectomy and Gastric Tube Reconstruction. Effect of Pneumatic Pylorus Dilatation During Hospital Stay, Surgical Complications During in Hospital Stay
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karolinska University Hospital (Other)
Collaborators: Lund University Hospital (Other); Sahlgrenska University Hospital (Other); Region Örebro County (Other); Uppsala University Hospital (Other); University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/896-31/4; 2013/896-31/4 (Other: Swedish Ethic Committee)
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Esophagectomy; No Signs of Cancer Recurrence; Delayed Gastric Emptying
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 15 mm Pyloric balloon dilatation. (Sham Comparator): During fluoroscopic control the pneumatic balloon is positioned of the pyloric sphincter and maintained there during the entire dilatation.
  Interventions: Other: 15 mm pyloric balloon dilatation
- Pneumatic pyloric dilatation. (Active Comparator): Endoscopy and 15 mm balloon dilatation is completed according to the same principle as active comparator arm.
  Interventions: Device: Pneumatic pyloric dilatation

INTERVENTIONS:
Device: Pneumatic pyloric dilatation
  Arms: Pneumatic pyloric dilatation.
Other: 15 mm pyloric balloon dilatation
  Arms: 15 mm Pyloric balloon dilatation.

SUMMARY:
Delayed emptying of the gastric tube after esophagectomy is a frequent and durable problem. No treatment is currently available. It can be hypothesized that incomplete relaxation of the pyloric sphincter may be a significant contributing factor. Pneumatic dilatation may therefore be a potentially effective treatment.

DETAILED DESCRIPTION:
Patients surviving one year after esophagectomy are sent questionnaires to pick up symptoms suggestive of delayed gastric emptying.Those fulfilling predefined criteria for delayed gastric emptying will be invited to the study. The study design is sham controlled single blind with a follow up extending to twelve months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previous esophagectomy and gastric tube reconstruction.
* Symptoms suggestive of delayed gastric emptying.
* signed informed consent

Exclusion Criteria:

* Signs of recurrent cancer disease
* no symptoms suggestive of delayed gastric emptying.
* unwillingness to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms suggestive of delayed gastric emptying | 3-12 months after treatment
  Symptoms will be assessed at 3, 6 and 12 months after therapy. In case of failure the code will be broken and if sham procedure has been done the patient will be offered pneumatic dilatation.

SECONDARY OUTCOMES:
Quality of Life | 3-12 months after treatment.
  Symptoms will be assessed at 3, 6 and 12 months after therapy. In case of failure the code will be broken and if sham procedure has been done the patient will be offered pneumatic dilatation.
Delayed gastric emptying | 3, 6 and 12 months after treatment.
  Symptoms will be assessed at 3, 6 and 12 months after therapy. In case of failure the code will be broken and if sham procedure has been done the patient will be offered pneumatic dilatation. Paracetamol test done only 3 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Tsai, ass professor, Principal Investigator — Karolinska University Hospital, Gastrocentrum
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden